CLINICAL TRIAL: NCT01661283
Title: Phase 2 Study of the mTOR Inhibitor Everolimus in Combination With Bevacizumab in Patients With Sporadic and Neurofibromatosis Type 1 (NF1) Related Refractory Malignant Peripheral Nerve Sheath Tumors
Brief Title: SARC016: Study of Everolimus With Bevacizumab to Treat Refractory Malignant Peripheral Nerve Sheath Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Genentech, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC016
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Malignant Peripheral Nerve Sheath Tumors; MPNST; Sarcoma
Keywords: MPNST; malignant peripheral nerve sheath tumors; RAD001; Everolimus; Bevacizumab; Sarcoma; Avastin; mTOR inhibitor
MeSH Terms: conditions — Neurofibrosarcoma; Sarcoma | interventions — Everolimus; Bevacizumab

ARMS (1):
- Arm A (Experimental): All patients with MPNST will continue everolimus 10 mg daily and bevacizumab 10 mg/kg dose every 14 days
  Interventions: Drug: everolimus; Drug: bevacizumab

INTERVENTIONS:
Drug: everolimus — 10 mg tablet once daily
  Other Names: Afinitor, everolimus
Drug: bevacizumab — 10 mg/kg dose every 14 days
  Other Names: Avastin

SUMMARY:
To determine the clinical response rate of everolimus in combination with bevacizumab for patients with chemotherapy refractory sporadic or neurofibromatosis type 1 (NF1) associated malignant peripheral nerve sheath tumor (MPNST). To evaluate the toxicity and safety of everolimus in combination with bevacizumab in individuals with MPNST

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 or older
* Unresectable or metastatic sporadic or NF1 associated high-grade MPNST
* Experienced progression after one or more prior regimens of cytotoxic chemotherapy
* Patients must be able to swallow tablets
* Patients must have measurable disease, defined as at least one tumor that is measurable
* Patients who develop a recurrence or progression (WHO criteria) of an MPNST in a previously radiated field may be enrolled if it has been at least 4 weeks since the last dose of radiation therapy
* Patients must have recovered from the toxic effects of all prior therapy before entering this study
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patents who received an anthracycline prior to enrollment must have an ejection fraction ≥ 50%
* Subjects of childbearing potential requires acceptable form of birth control
* Informed consent

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 3 weeks of the start of study drug or patients receiving prior treatment with investigational drugs 4 weeks of the start of study drug
* Patients may not be currently receiving strong inhibitors of CYP3A4, and may not have received these medications within 1 week of entry
* Prior radiotherapy within 4 weeks of the start of study drug
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug,
* Patients who have not recovered from the side effects of any major surgery
* Patients that may require major surgery during the course of the study
* Less than 7 days have passed from core biopsies or other minor surgical procedures excluding placement of a vascular access device
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent(Topical or inhaled corticosteroids are allowed)
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Female patients who are pregnant or breast feeding
* Patients who have received prior treatment with an mTOR inhibitor or bevacizumab
* Patients with known hypersensitivity to rapamycins
* concurrent use of anti-coagulant drugs
* Patients using Seville orange, star fruit, grapefruit and their juices, and St. John's Wort
* Patients taking enzyme inducing anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-09; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C. Widemann, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania

REFERENCES:
- See also: SARC Website — http://www.sarctrials.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Everolimus (2.5, 5, and 10 mg tablets) was administered at 10 mg per dose once daily at the same time on a continuous dosing schedule.
  Bevacizumab (400 mg vials) was administered at 10 mg/kg as intravenous infusion over 30-90 minutes every 2 weeks (days 1 and 15).
  One treatment cycle was 28 days.
Period: Overall Study
Arm/Group | Treatment
Started | 25 (15 patients enrolled in the first stage; 10 patients enrolled in the second stage)
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 17 patients enrolled with NF1 and 8 patients enrolled with sporadic MPNST.
Arm/Group | Treatment
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] — Population: 17 patients enrolled with NF1 and 8 patients enrolled with sporadic MPNST.
  years
    All | 37 [19 to 81]
    NF1: number analyzed (Participants) | 17
    NF1 | 28 [19 to 63]
    Sporadic: number analyzed (Participants) | 8
    Sporadic | 61 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Was the primary tumor resected [Count of Participants; unit: Participants]
  No | 5
  Yes | 20
Patient had prior chemotherapy [Count of Participants; unit: Participants]
  No | 2
  Yes | 23
Patient had prior radiation [Count of Participants; unit: Participants]
  No | 4
  Yes | 21
ECOG performance score at baseline [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Scale:
  Grade 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature.
  Grade 2: In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 12
    1 | 11
    2 | 2
Margins of surgical resection [Count of Participants; unit: Participants] — Population: 20 subjects had the primary tumor resected out of the 25 total subjects.
  Participants
    number analyzed (Participants) | 20
    Unknown | 2
    R0- All Margins Pathologically Negative | 9
    R1- Microscopically Positive Margins | 4
    R2- Macroscopically Positive Margins | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (Complete Response, Partial Response, and Stable Disease at ≥ 4 Months Using World Health Organization (WHO) Criteria) of Everolimus in Combination With Bevacizumab
Description: Evaluate if the combination of the mTOR inhibitor everolimus combined with the angiogenesis inhibitor bevacizumab would result in a modest clinical benefit rate, which included confirmed partial and complete responses and disease stability for four or more treatment cycles based on WHO Response Criteria. Per WHO for target lesions: Complete Response (CR): Disappearance of all known disease, determined by two consecutive observations not less than 4 weeks apart.
  Partial Response (PR): A > 50% decrease in the total tumor load of the lesions that have been measured to determine the effect of therapy not less than four weeks apart. The observations must be consecutive. Stable Disease (SD): A 50% decrease in total tumor area cannot be established nor has a 25% increase in the size of one or more measurable lesions been demonstrated.
Time Frame: Assessed at Baseline and prior to Cycle 3, 5, 7, 9, etc., for up to 2 years. 1 cycle =28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 25
Participants | 3

2. Secondary Outcome: Spectrum of Germline NF1 Mutations in Individuals With NF1 Associated MPNSTs
Description: To evaluate the spectrum of germline NF1 mutations in individuals with NF1 associated MPNSTs
Time Frame: greater than or equal to 4 months
Population: NF1 germline mutations were not analyzed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Response Stratified by Individuals With Sporadic or NF1 Associated MPNST
Description: To explore differences in the response rate to everolimus in combination with bevacizumab in individuals with sporadic and NF1 associated MPNST. Responses include confirmed partial and complete responses and disease stability for four or more treatment cycles based on WHO Response Criteria. Per WHO for target lesions: Complete Response (CR): Disappearance of all known disease, determined by two consecutive observations not less than 4 weeks apart. Partial Response (PR): A > 50% decrease in the total tumor load of the lesions that have been measured to determine the effect of therapy not less than four weeks apart. The observations must be consecutive. Stable Disease (SD): A 50% decrease in total tumor area cannot be established nor has a 25% increase in the size of one or more measurable lesions been demonstrated.
Time Frame: Assessed at Baseline and prior to Cycle 3, 5, 7, 9, etc., for up to 2 years. 1 cycle =28 days
Population: The rows are broken up by patients with NF1 associated MPNST (n=17) and sporadic MPNST (n=8)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 25
Participants
  NF1 associated MPNST: number analyzed (Participants) | 17
  NF1 associated MPNST | 2
  Sporadic MPNST: number analyzed (Participants) | 8
  Sporadic MPNST | 1

4. Secondary Outcome: Relationship Between Response to Everolimus in Combination With Bevacizumab and the Presence of NF1 Mutations or NF1 Inactivation in MPNST Tumor Samples
Description: To explore the relationship between response to everolimus in combination with bevacizumab and the presence of NF1 mutations or NF1 inactivation in MPNST tumor samples
Time Frame: greater than or equal to 4 months
Population: Tumor samples were not analyzed for NF1 mutations.
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Vascular Endothelial Growth Factor (VEGF) and Vascular Endothelial Growth Factor Receptor 2 (VEGFR2) Levels at Baseline and Pre-Cycles 3 and 5
Description: To assess changes in Vascular Endothelial Growth Factor (VEGF) and Vascular Endothelial Growth Factor Receptor 2 (VEGFR2) Levels in peripheral blood specimens during treatment.
Time Frame: Baseline, Pre-Cycle 3, Pre-Cycle 5
Population: Paired samples for analysis were collected for 14 patients at baseline and time of first restaging and 8 patients at time of second restaging.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Treatment
Number analyzed (Participants) | 14
pg/mL
  VEGF- Baseline | 103.58 [31.20 to 593.61]
  VEGF- Pre Cycle 3 | 184.24 [55.82 to 334.49]
  VEGF- Pre Cycle 5: number analyzed (Participants) | 8
  VEGF- Pre Cycle 5 | 192.49 [138.51 to 262.94]
  VEGFR2- Baseline | 1363.76 [1043.25 to 2109.18]
  VEGFR2 Pre Cycle 3 | 911.89 [658.63 to 1815.49]
  VEGFR2 Pre Cycle 5: number analyzed (Participants) | 8
  VEGFR2 Pre Cycle 5 | 863.85 [500.85 to 1678.16]

6. Secondary Outcome: Utility of 3-D MRI Analysis in Comparison to 1-D and 2-D Measurements to More Sensitively Monitor Response to Everolimus in Combination With Bevacizumab
Description: To evaluate the utility of 3-D MRI analysis in comparison to 1-D and 2-D measurements to more sensitively monitor response to everolimus in combination with bevacizumab
Time Frame: greater than or equal to 4 months
Population: Imaging studies of sufficient quality to analyze tumors were not collected. Therefore, unable to analyze volumes and compare 3-D to 1-D and 2-D measurements.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: ~4 years
Description: CTCAE version 4.0
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Death NOS (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=25)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Platelet count decreased (Blood and lymphatic system disorders) | 4 (6)
White blood cell decreased (Blood and lymphatic system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 12 (20)
Oral pain (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 5 (6)
Fever (General disorders) | 2 (2)
Fatigue (General disorders) | 11 (14)
Alanine aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Weight loss (Investigations) | 8 (9)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Cholesterol high (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (10)
Muscle weakness (lower limb, upper limb) (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)
Pain (neck, back, chest wall, ear, flank) (General disorders) | 5 (7)
Insomnia (Psychiatric disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT01661283/Prot_SAP_000.pdf